CLINICAL TRIAL: NCT04813731
Title: COVID-19 And Lingering Symptoms In Primary Care Patients
Acronym: CALIP
Status: Completed | Type: Observational
Sponsor: Katarina Hedin (Other Government)
Collaborators: Research Unit for General Practice in Aalborg (Other); Utrecht University (Other); National University of Ireland, Galway, Ireland (Other); Region Jönköping County (Other Government)
Responsible Party: Sponsor-Investigator, Katarina Hedin, Adjunct professor, Region Jönköping County
Organization: Region Jönköping County (Other Government)
Other Study IDs: 2020-05448
Record Dates: First submitted 2021-03-07; First posted 2021-03-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Covid19; Symptoms and Signs
MeSH Terms: conditions — COVID-19; Signs and Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The ongoing corona virus disease 2019 (COVID-19) is a viral acute respiratory tract infection caused by server acute respiratory syndrom coronavirus typ 2 (SARS-CoV-2). The signs and symptom of SARS-CoV-2 infection vary and most people with COVID-19 experience illness of mild or moderate severity and recover with symptomatic treatment outside of hospital. Studies have found that some people experience lingering/long-lasting symptoms and only a minority of patients were completely free from COVID-19 related symptoms after two months. About one third still had up to two residual symptoms and 55% had three or more. As far as we know no study on lingering symptoms has been published in patients after a mild or moderate infection managed in primary care settings. The aim of this study is to explore the course of disease over a one year period and describe lingering symptoms and their impact on well-being and daily activities in adult non-hospitalized patients with previous established COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed SARS-CoV-2 infection, either by polymeras chain reaction (PCR), or by antigen testing (if authorized/recommended/used by national/local governments)
* Symptoms consistent with mild to moderate COVID-19
* Maximum of 2 weeks since positive SARS-CoV-2 test
* Aged 18 years and older
* Patient able and willing to comply with monthly phone calls.

Exclusion Criteria:

* Hospitalisation due to COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients over all age categories with laboratory confirmed SARS-CoV-2 infection and symptoms consistent with COVID-19
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Time to full recovery symptoms | through study completion, a maximum of 1 year
  Number of weeks until "back to normal"

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Hedin, Assoc Prof, Principal Investigator — Region Jönköping County Sweden
Locations (13):
- Belgium (2):
  - Centre for General Practice, Department of Family Medicine & Population Health (FAMPOP), Faculty of Medicine and Health Sciences, University of Antwerp, Antwerp
  - the Academic Centre for General Practice (ACHG), Department of Public Health and Primary Care, KU Leuven, Leuven
- Center for General Practice at Aalborg University, Aalborg, Denmark
- Département de Santé Publique, Université Côte d'Azur, Centre Hospitalier Universitaire de Nice, Nice, France, Nice, France
- R. Lugar Center for Public Health Research, Tbilisi, Georgia
- Institut für Allgemeinmedizin Universitätsklinikum Würzburg Josef-Schneider-Str. 2/D7 97080 Würzburg, Würzburg, Germany
- School of Medicine, National University of Ireland, Galway, Ireland
- Covid-19 primary care special unit Sassuolo, Azienda Unità Sanitaria locale di Modena, Modena, Italy, Modena, Italy
- Julius Center, University Medical Center Utrecht, Utrecht, Netherlands
- Medical University of Lodz, Lodz, Lodz, Poland
- Balan Medfam SRL, Cluj-Napoca, Romania
- Sweden (2):
  - Wetterhälsan Primary Health Care Centre, Jönköping
  - Kärna Primary Health Care Centre, Linköping

IPD SHARING:
Plan to Share IPD: No